CLINICAL TRIAL: NCT01755949
Title: Impact and Time Course of Colchicine Therapy on C-reactive Protein Elevation in Chronic Atrial Fibrillation (AF) and Post AF Ablation
Brief Title: Colchicine and CRP in Atrial Fibrillation and AF Ablation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Takeda (Industry); Detiger Funds (Unknown)
Responsible Party: Principal Investigator, Joseph L. Blackshear, Principal Investiator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-001686
Record Dates: First submitted 2012-12-19; First posted 2012-12-24 (Estimated); Results first posted 2019-05-09 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-04

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; catheter ablation; colchicine; c reactive protein; CRP
MeSH Terms: conditions — Atrial Fibrillation | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Chronic atrial fibrillation, colchicine (Active Comparator): Colchicine 0.6 mg PO BID. Subjects not undergoing ablation.
  Interventions: Drug: Colchicine, 0.6 mg PO BID
- Chronic atrial fibrillation, placebo (Placebo Comparator): Matching placebo. Subjects not undergoing ablation.
  Interventions: Drug: Matching placebo
- Pre-ablation, sinus rhythm, colchicine (Active Comparator): Colchicine 0.6 mg PO BID. Subjects undergoing ablation.
  Interventions: Drug: Colchicine, 0.6 mg PO BID
- Pre-ablation, sinus rhythm, placebo (Placebo Comparator): Matching placebo. Subjects undergoing ablation.
  Interventions: Drug: Matching placebo
- Pre-ablation, AF, colchicine (Active Comparator): Colchicine 0.6 mg PO BID. Subjects undergoing ablation.
  Interventions: Drug: Colchicine, 0.6 mg PO BID
- Pre-ablation, AF, placebo (Placebo Comparator): Matching placebo. Subjects undergoing ablation.
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Colchicine, 0.6 mg PO BID — Colchicine tablets will be over-encapsulated by the research pharmacy to be indistinguishable from placebo
  Other Names: Colcrys
  Arms: Chronic atrial fibrillation, colchicine; Pre-ablation, AF, colchicine; Pre-ablation, sinus rhythm, colchicine
Drug: Matching placebo — Matching placebo tablets will be encapsulated by the research pharmacy to be indistinguishable from active drug
  Other Names: placebo
  Arms: Chronic atrial fibrillation, placebo; Pre-ablation, AF, placebo; Pre-ablation, sinus rhythm, placebo

SUMMARY:
Colchicine will lower C-reactive protein (CRP) in chronic atrial fibrillation and reduce the rise in CRP which occurs following atrial fibrillation ablation

DETAILED DESCRIPTION:
Three groups of patients will be randomized to colchicine 0.6 mg PO bis in die (BID) or matching placebo:

1. Paroxysmal atrial fibrillation, pre-ablation
2. Persistent atrial fibrillation, pre-ablation
3. Chronic persistent atrial fibrillation

ELIGIBILITY:
Inclusion Criteria:

* Group 1: Persistent or chronic AF presenting for evaluation in cardiology offices. Diagnosis of AF will be made based on the 12 -lead surface ECG.
* Group 2: Paroxysmal AF scheduled to go AF ablation presenting to the electrophysiology laboratory for the procedure in sinus rhythm..
* Group 3:Chronic AF scheduled to go clinically indicated AF ablation, and presenting in the electrophysiology laboratory in atrial fibrillation .

Exclusion Criteria:

1. Abnormal liver function with elevated enzymes> 1.5 times the normal.
2. Abnormal kidney function with glomerular filtration rate < 50 ml/min
3. Increased levels of creatine kinase or known myopathy
4. Neutropenia
5. Known GI disorders
6. Women of childbearing age who have not had surgical sterilization and are not using oral contraceptives, or who's spouse has not had surgical sterilization will be excluded due to the length of the trial and the possibility that they could become pregnant after entry.
7. Pregnant and lactating women
8. Lactose intolerance
9. Known sensitivity, allergy, or contraindication to colchicine use

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-03; Primary Completion 2016-12-06 (Actual); Study Completion 2016-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph L. Blackshear, MD, Principal Investigator — Consultant in Cardiovascular Diseases
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Chronic Atrial Fibrillation, Colchicine: Colchicine 0.6 mg PO bis in die (BID)
  Colchicine, 0.6 mg PO BID: Colchicine tablets will be over-encapsulated by the research pharmacy to be indistinguishable from placebo
  Subjects not undergoing ablation.
- Chronic Atrial Fibrillation, Placebo: Matching placebo
  Matching placebo: Matching placebo tablets will be encapsulated by the research pharmacy to be indistinguishable from active drug
  Subjects not undergoing ablation.
- Pre-ablation, Sinus Rhythm, Colchicine; Pre-ablation, AF, Colchicine: Colchicine 0.6 mg PO BID
  Colchicine, 0.6 mg PO BID: Colchicine tablets will be over-encapsulated by the research pharmacy to be indistinguishable from placebo Subjects undergoing ablation.
- Pre-ablation, Sinus Rhythm, Placebo; Pre-ablation, AF, Placebo: Matching placebo
  Matching placebo: Matching placebo tablets will be encapsulated by the research pharmacy to be indistinguishable from active drug
  Subjects undergoing ablation.
Period: Overall Study
Arm/Group | Chronic Atrial Fibrillation, Colchicine | Chronic Atrial Fibrillation, Placebo | Pre-ablation, Sinus Rhythm, Colchicine | Pre-ablation, Sinus Rhythm, Placebo | Pre-ablation, AF, Colchicine | Pre-ablation, AF, Placebo
Started | 5 | 5 | 4 | 5 | 4 | 3
Completed | 5 | 5 | 4 | 5 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Chronic Atrial Fibrillation, Colchicine: Colchicine 0.6 mg PO BID
  Colchicine, 0.6 mg PO BID: Colchicine tablets will be over-encapsulated by the research pharmacy to be indistinguishable from placebo Subjects not undergoing ablation.
- Total: Total of all reporting groups
Arm/Group | Chronic Atrial Fibrillation, Colchicine | Chronic Atrial Fibrillation, Placebo | Pre-ablation, Sinus Rhythm, Colchicine | Pre-ablation, Sinus Rhythm, Placebo | Pre-ablation, AF, Colchicine | Pre-ablation, AF, Placebo | Total
Number analyzed (Participants) | 5 | 5 | 4 | 5 | 4 | 3 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (7) | 73 (8) | 65 (5) | 69 (6) | 68 (7) | 62 (18) | 68 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 1 | 0 | 0 | 4
  Male | 3 | 4 | 4 | 4 | 4 | 3 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 5 | 4 | 4 | 5 | 4 | 3 | 25
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 4 | 5 | 4 | 3 | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in C-reactive Protein
Description: Plasma levels of C-reactive protein was determined by the immunoprecipitation method using an in vitro diagnostic assay.
Time Frame: baseline, day 28
Population: Not all subjects had sample available at all timepoints to measure C-reactive protein levels. Sample was either not collected or insufficient volume to run assay.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Chronic Atrial Fibrillation, Colchicine: Colchicine 0.6 mg, twice daily for 28 days Subjects not undergoing ablation.
- Chronic Atrial Fibrillation, Placebo: Placebo tablets, encapsulated to be indistinguishable from active drug, twice daily for 28 days Subjects not undergoing ablation.
- Pre-ablation, Sinus Rhythm, Colchicine; Pre-ablation, AF, Colchicine: Colchicine 0.6 mg, twice daily for 28 days Subjects undergoing ablation.
- Pre-ablation, Sinus Rhythm, Placebo; Pre-ablation, AF, Placebo: Placebo tablets, encapsulated to be indistinguishable from active drug, twice daily for 28 days Subjects undergoing ablation.
Arm/Group | Chronic Atrial Fibrillation, Colchicine | Chronic Atrial Fibrillation, Placebo | Pre-ablation, Sinus Rhythm, Colchicine | Pre-ablation, Sinus Rhythm, Placebo | Pre-ablation, AF, Colchicine | Pre-ablation, AF, Placebo
Number analyzed (Participants) | 5 | 5 | 4 | 5 | 3 | 3
ng/mL
  Baseline | 6.4 (7.2) | 2.7 (2.9) | 2.9 (1.6) | 5.9 (5.5) | 2.6 (2.7) | 2.3 (1.7)
  day 28: number analyzed (Participants) | 5 | 5 | 2 | 4 | 3 | 2
  day 28 | 1.8 (2.0) | 2.7 (1.4) | 1.0 (0.7) | 2.5 (1.7) | 1.2 (1.0) | 5.2 (5.1)
Statistical Analysis 1: Comparison: Chronic Atrial Fibrillation, Colchicine vs Pre-ablation, Sinus Rhythm, Colchicine vs Pre-ablation, AF, Colchicine; Baseline C-reactive protein vs day 28 C-reactive protein; Test type: Superiority; p = 0.038, t-test, 2 sided
Statistical Analysis 2: Comparison: Chronic Atrial Fibrillation, Placebo vs Pre-ablation, Sinus Rhythm, Placebo vs Pre-ablation, AF, Placebo; Baseline C-reactive protein vs day 28 C-reactive protein; Test type: Superiority; p = 0.98, t-test, 2 sided
Statistical Analysis 3: Comparison: Chronic Atrial Fibrillation, Colchicine vs Chronic Atrial Fibrillation, Placebo vs Pre-ablation, Sinus Rhythm, Colchicine vs Pre-ablation, Sinus Rhythm, Placebo vs Pre-ablation, AF, Colchicine vs Pre-ablation, AF, Placebo; difference between placebo and colchicine levels at day 28; Test type: Superiority; p = 0.072, t-test, 2 sided

2. Secondary Outcome: Number of Subjects With Atrial Fibrillation
Description: All subjects will have 12 lead ECG on day 28 to measure the number of subjects with normal sinus rhythm and atrial fibrillation.
Time Frame: day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic Atrial Fibrillation, Colchicine | Chronic Atrial Fibrillation, Placebo | Pre-ablation, Sinus Rhythm, Colchicine | Pre-ablation, Sinus Rhythm, Placebo | Pre-ablation, AF, Colchicine | Pre-ablation, AF, Placebo
Number analyzed (Participants) | 5 | 5 | 4 | 4 | 4 | 3
Participants
  Sinus rhythm | 5 | 1 | 4 | 3 | 4 | 1
  Atrial fibrillation | 0 | 4 | 0 | 1 | 0 | 2
Statistical Analysis 1: Comparison: Chronic Atrial Fibrillation, Colchicine vs Pre-ablation, Sinus Rhythm, Colchicine vs Pre-ablation, Sinus Rhythm, Placebo vs Pre-ablation, AF, Colchicine vs Pre-ablation, AF, Placebo; placebo vs colchicine; Test type: Superiority; p = 0.08, t-test, 2 sided

3. Secondary Outcome: Time Course of C-reactive Protein Levels
Description: Plasma levels of C-reactive protein was determined by the immunoprecipitation method using an in vitro diagnostic assay.
Time Frame: baseline, day 3, day 7, day 14, day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Chronic Atrial Fibrillation, Colchicine | Chronic Atrial Fibrillation, Placebo | Pre-ablation, Sinus Rhythm, Colchicine | Pre-ablation, Sinus Rhythm, Placebo | Pre-ablation, AF, Colchicine | Pre-ablation, AF, Placebo
Number analyzed (Participants) | 5 | 5 | 4 | 5 | 4 | 3
ng/ml
  Baseline | 6.4 (7.2) | 2.7 (2.9) | 2.9 (1.6) | 5.9 (5.5) | 2.6 (2.7) | 2.3 (1.7)
  Day 3: number analyzed (Participants) | 5 | 5 | 3 | 3 | 3 | 2
  Day 3 | 4.3 (5.1) | 2.9 (2.2) | 24.9 (19.5) | 27.8 (2.82) | 4.4 (1.1) | 48.2 (59.0)
  Day 7: number analyzed (Participants) | 5 | 5 | 3 | 4 | 3 | 3
  Day 7 | 3.2 (4.8) | 3.2 (2.2) | 5.0 (2.2) | 6.6 (5.8) | 1.9 (1.2) | 15.4 (17.1)
  Day 14: number analyzed (Participants) | 5 | 5 | 3 | 4 | 3 | 2
  Day 14 | 4.3 (7.8) | 3.2 (2.3) | 1.9 (1.2) | 4.1 (3.0) | 2.0 (1.9) | 5.3 (0.9)
  Day 28: number analyzed (Participants) | 5 | 5 | 2 | 4 | 3 | 2
  Day 28 | 1.8 (2.0) | 2.7 (1.4) | 1.0 (0.7) | 2.5 (1.7) | 1.2 (1.0) | 5.2 (5.1)

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Chronic Atrial Fibrillation, Colchicine | Chronic Atrial Fibrillation, Placebo | Pre-ablation, Sinus Rhythm, Colchicine | Pre-ablation, Sinus Rhythm, Placebo | Pre-ablation, AF, Colchicine | Pre-ablation, AF, Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/4 | 0/5 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/4 | 0/5 | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/4 | 0/5 | 0/4 | 0/3

LIMITATIONS AND CAVEATS:
Enrollment was halted in 2015 due to departure of study staff; shortly thereafter Takeda Inc announced it could not renew production of colchicine nor support the study after the end of 2016. Principal investigator elected to terminate enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes